CLINICAL TRIAL: NCT00141947
Title: Safety and Efficacy of Add-On Oral Bexarotene to Antipsychotic Treatment in Schizophrenia Patients: An Open Label Trial
Brief Title: Bexarotene Treatment in Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Vladimir Lerner, Associated Professor, Beersheva Mental Health Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMHC-3775
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2005-10

CONDITIONS: Schizophrenia
Keywords: bexarotene; schizophrenia; psychopathology; cognitive impairment; quality of life; open lable trial
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bexarotene (Targretin)

SUMMARY:
In this proposed study, we aim to investigate the effects of Bexarotene (Targretin; LGD1069; 4-[1-{5,6,7,8-tetrahydro-3,5,5,8,8-pentamethyl-2-naphthalenyl} ethenyl] benzoic acid) on severity of psychopathology, cognitive impairment, and quality of life in schizophrenia patients in an open label trial. The rationale behind add-on oral bexarotene to ongoing antipsychotic treatment in schizophrenia patients is based on both the retinoid dysregulation hypothesis (Goodman, 1995) and the growth factors deficiency and synaptic destabilization hypothesis (Moises et al, 2002) of schizophrenia. In this clinical trial, a novel regimen of low dose bexarotene (Targretin, 75 mg/day) will be added for 6 weeks to the standard treatment of 15 schizophrenia patients on stable antipsychotic treatment. Participants will be assessed at baseline and after 2, 4 and 6 weeks of treatment. A battery of research instruments will be used for assessment of efficacy and safety (psychopathology, and side effects). In addition, cholesterol and triglyceride levels, liver and thyroid function tests and a blood cell count will be monitored at baseline and during therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60
* schizophrenia
* stable blood parameters
* normal baseline fasting triglyceride
* ability to sign informed consent

Exclusion Criteria:

* lipid abnormalities
* leukopenia or neutropenia
* organic brain damage (mental retardation)
* alcohol or drug abuse
* renal disease
* hepatic dysfunction
* history of pancreatitis
* thyroid axis alterations
* suicide attempt in past year
* cataracts
* systemic treatment with more than 15,000IU vitamin A daily
* patients with known hypersensitivity to bexarotene or other components of the product
* pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Schedule for Assessment of Mental Disorder
The Positive and Negative Syndrome Scale
Montgomery and Äsberg Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev; Michael Ritsner, MD, Principal Investigator — Technion-Israel Institute of Technology (Haifa)
Locations (2):
- Israel (2):
  - Beersheva Mental Health Center, Beersheva
  - Shaar Manashe Mental Health Center, Hadera

REFERENCES:
- [Derived] Lerner V, Miodownik C, Gibel A, Kovalyonok E, Shleifer T, Goodman AB, Ritsner MS. Bexarotene as add-on to antipsychotic treatment in schizophrenia patients: a pilot open-label trial. Clin Neuropharmacol. 2008 Jan-Feb;31(1):25-33. doi: 10.1097/WNF.0b013e31806450da. PMID 18303488